CLINICAL TRIAL: NCT05453110
Title: Does Self-efficacy Predict Outcomes Among U.S. Military Academy Cadets During Initial Entry Training?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KACH.2022.0053
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Low Back Pain; Musculoskeletal Injury
Keywords: Nocebo; Self-Efficacy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Group Between-Factor, Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cautionary (Experimental): The group will receive a message regarding potential risk for spine injury before the tested task.
  Interventions: Behavioral: Deadlift Form Education
- Reassuring (Experimental): This group will receive a message regarding spine resiliency before the tested task.
  Interventions: Behavioral: Deadlift Form Education
- Control (No Intervention): This group will not receive education before the tested task.

INTERVENTIONS:
Behavioral: Deadlift Form Education — The education will include information about the lumbar spine as it relates to a deadlift. The researchers will administer this education shortly prior to participants taking a strength test.
  Arms: Cautionary; Reassuring

SUMMARY:
Background:

Lower back injuries are a common occurrence in athletes, sports programs, and in the military (Bengtsson, 2018; Lovalekar, 2021). The Army's new fitness test includes a three-repetition maximum deadlift, and this inclusion has raised concern amongst servicemembers and healthcare workers due to the association between deadlifts and lower back injuries. There is debate amongst researchers about the role of deadlift form in lower back injury prevention, specifically related to flexion of the spine (Sjoberg, 2020).

Purpose:

The purpose of this study is to investigate the effect of low back pain education (either cautionary regarding injury risk or reassuring regarding spine resiliency) on deadlift performance (weight lifted), and if this education has an effect on self-efficacy and perceived spine vulnerability.

Participants:

Participants will be incoming new cadets at the United States Military Academy (USMA). Inclusion criteria are cadets age 17-26 (cadets under the age of 18 are legally emancipated therefore able to consent), those participating in the ACFT, and speak and understand English.

Study Design:

This study will be a randomized controlled trial with parallel design and 1:1 allocation ratio. The investigators plan to use cluster randomization. There will be three groups- control, cautionary, reassuring (Jackson, 2005). The investigators are also planning a prospective cohort study to assess self-efficacy, injury, and performance over time.

Procedures:

Data will be collected at the United States Military Academy during the summer of 2022 during cadet basic training. Shortly after new cadets arrive at USMA, the investigators will gather demographic and initial self-efficacy information. The randomized control element of this study will occur before and during the maximum deadlift (MDL) of the Army Combat Fitness Test (ACFT). At the start of cadet basic training, investigators will randomly allocate each company of cadets into one of three groups (three companies per group.) The investigator will administer the education (cautionary, reassuring, or control) shortly prior to cadets taking the MDL, and will collect results after the ACFT. The cautionary education is similar to standard information provided to many servicemembers before the start of an ACFT or a maximum deadlift.

DETAILED DESCRIPTION:
Background:

Musculoskeletal injuries (MSKIs) are the leading cause of nondeployability, lost duty days (LDD), medical encounters, military discharge, and disability in the United States Military. (Lovalekar, 2021). Ironically, the leading causes of MSKIs are same activities that leaders deliberately conduct to develop physical resilience: running, foot marching, other physical fitness training activities (besides running) and work-related tasks (Lovalekar, 2021).

Purpose:

The purpose of this study is to learn about relationships between self-efficacy, injury and physical/tactical performance. The investigators also plan to assess the effect of low back pain education (either cautionary regarding injury risk or reassuring regarding spine resiliency) on deadlift performance (weight lifted), and if this education has an effect on self-efficacy and perceived spine vulnerability.

Participants:

Participants will be incoming new cadets at the United States Military Academy (USMA). Inclusion criteria are cadets age 17-26 (cadets under the age of 18 are legally emancipated therefore able to consent), those participating in the ACFT, and speak and understand English.

Study Design:

This study will be a randomized controlled trial with parallel design and 1:1 allocation ratio. The investigators plan to use cluster randomization. There will be three groups- control, cautionary, reassuring (Jackson, 2005). The investigators are also planning a prospective cohort study to assess self-efficacy, injury, and performance over time.

Procedures:

Data will be collected at the United States Military Academy during the summer of 2022 during cadet basic training. Shortly after new cadets arrive at USMA, the investigators will gather demographic and initial self-efficacy information. The randomized control element of this study will occur before and during the maximum deadlift (MDL) of the Army Combat Fitness Test (ACFT). At the start of cadet basic training, researchers will randomly allocate each company of cadets into one of three groups (three companies per group.) The researchers will administer the education (cautionary, reassuring, or control) shortly prior to cadets taking the MDL, and will collect results after the ACFT. The cautionary education is similar to standard information provided to many servicemembers before the start of an ACFT or a maximum deadlift.

ELIGIBILITY:
Inclusion Criteria:

* All incoming US Military Academy cadets, attending cadet basic training in summer 2022.

Exclusion Criteria:

* Unable to communicate in English; unable to participate in deadlift event.

Ages: 17 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 903 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Keller Army Community Hospital, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jackson T, Pope L, Nagasaka T, Fritch A, Iezzi T, Chen H. The impact of threatening information about pain on coping and pain tolerance. Br J Health Psychol. 2005 Sep;10(Pt 3):441-51. doi: 10.1348/135910705X27587. PMID 16238858
- [Result] Bengtsson V, Berglund L, Aasa U. Narrative review of injuries in powerlifting with special reference to their association to the squat, bench press and deadlift. BMJ Open Sport Exerc Med. 2018 Jul 17;4(1):e000382. doi: 10.1136/bmjsem-2018-000382. eCollection 2018. PMID 30057777
- [Result] Lovalekar M, Hauret K, Roy T, Taylor K, Blacker SD, Newman P, Yanovich R, Fleischmann C, Nindl BC, Jones B, Canham-Chervak M. Musculoskeletal injuries in military personnel-Descriptive epidemiology, risk factor identification, and prevention. J Sci Med Sport. 2021 Oct;24(10):963-969. doi: 10.1016/j.jsams.2021.03.016. Epub 2021 Mar 31. PMID 33824080
- [Result] Sjoberg H, Aasa U, Rosengren M, Berglund L. Content Validity Index and Reliability of a New Protocol for Evaluation of Lifting Technique in the Powerlifting Squat and Deadlift. J Strength Cond Res. 2020 Sep;34(9):2528-2536. doi: 10.1519/JSC.0000000000002791. PMID 30199449
- [Derived] Scott KM, Kreisel BR, Florkiewicz EM, Crowell MS, Morris JB, McHenry PA, Benedict TM. The Effect of Cautionary Versus Resiliency Spine Education on Maximum Deadlift Performance and Back Beliefs: A Randomized Control Trial. J Strength Cond Res. 2024 Jul 1;38(7):e341-e348. doi: 10.1519/JSC.0000000000004783. Epub 2024 May 28. PMID 38900182

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 903 new cadets consented to the study and signed informed consent forms. 18 of them were separated from the academy before data collection, and 64 were injured prior to data collection and did not take the fitness test. Of the 64 participants who were injured, 16 received the intervention but did not take the fitness test, thus we did not collect primary outcome data. This resulted in 837 who received the intervention. There were 821 participants who were included in the final analysis.
Period: Overall Study
Arm/Group | Cautionary | Reassuring | Control
Started (Individuals who received the intervention) | 269 | 283 | 285
Completed | 264 | 278 | 279
Not Completed | 5 | 5 | 6
Not completed — Received intervention but did not complete primary outcome measure | 5 | 5 | 6

BASELINE CHARACTERISTICS:
Population: Includes all participants who consented to participate, including those who did not receive the intervention due to separation from the academy or injury prior to data collection. Because those participants consented and completed demographic and deadlift self-efficacy information before their separation/injury, we still included them as Baseline participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cautionary | Reassuring | Control | Total
Number analyzed (Participants) | 293 | 298 | 312 | 903
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.3 (1) | 18.2 (.9) | 18.3 (.9) | 18.3 (.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 63 | 73 | 198
  Male | 231 | 235 | 239 | 705
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kilograms] | 74.7 (13.3) | 74.3 (12.8) | 74.1 (11.7) | 74.4 (12.6)
Intercollegiate Athlete [Count of Participants; unit: Participants] | 101 | 89 | 96 | 286
Prior history of deadlift-related low back pain [Count of Participants; unit: Participants] | 30 | 37 | 49 | 116
Prior Military Service [Count of Participants; unit: Participants] | 52 | 47 | 54 | 153

OUTCOME MEASURES:

1. Primary Outcome: Maximum Deadlift Weight Lifted
Description: Weight lifted for three repetitions
Time Frame: Following the intervention. This event/data collection took place at a single time point immediately following the intervention, up to 30 minutes
Population: Includes only those who completed the primary outcome measure
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Cautionary | Reassuring | Control
Number analyzed (Participants) | 264 | 278 | 279
kilograms | 117.2 (25.9) | 115.9 (26.6) | 119.0 (27.1)

2. Primary Outcome: Perceived Spine Vulnerability, Q1
Description: Ease of which participants believe the back can be injured, "it is easy to injure your back". Questions based on Back Pain Attitude Questionnaire, item 6. Count reflects the number of participants who selected "true"
Time Frame: Immediately after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Cautionary | Reassuring | Control
Number analyzed (Participants) | 264 | 278 | 279
Participants | 153 | 136 | 114

3. Primary Outcome: Perceived Spine Vulnerability, Q2
Description: Ease of which participants believe the back can be injured, "you could injure your back if you are not careful". Questions based on Back Pain Attitude Questionnaire, item 11. Count reflects the number of participants who selected "true"
Time Frame: Immediately after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Cautionary | Reassuring | Control
Number analyzed (Participants) | 264 | 278 | 279
Participants | 242 | 251 | 227

4. Secondary Outcome: Deadlift Self-Efficacy Questionnaire
Description: Self-efficacy related to the deadlift was gathered by a single numeric rating scale question. Participants were asked to rate their confidence in succeeding at the deadlift event, from "not confident at all - 0" to "fully confident - 10).
Time Frame: Outcome data was collected immediately following the intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cautionary | Reassuring | Control
Number analyzed (Participants) | 264 | 278 | 279
score on a scale | 10 [8 to 10] | 10 [8 to 10] | 9 [8 to 10]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Cautionary | Reassuring | Control
All-Cause Mortality (participants affected / at risk) | 0/269 | 0/283 | 0/279
Serious Adverse Events (participants affected / at risk) | 0/269 | 0/283 | 0/285
Other Adverse Events (participants affected / at risk) | 0/269 | 0/283 | 0/285

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT05453110/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT05453110/ICF_001.pdf